CLINICAL TRIAL: NCT00214136
Title: A Phase II Prostate Cancer Trial Treating Pelvic Lymph Nodes to High Dose Using Intensity Modulated Radiation Therapy
Brief Title: Intensity Modulated Radiation Therapy (IMRT) Radiotherapy for Treating Prostate Pelvic Nodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO04807; P01CA088960 (NIH); H-2004-0472 (Other: Institutional Review Board); NCI-2011-00947 (Registry Identifier: NCI Trial ID); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): prostate radiation to 70Gy, lymph nodes to 56Gy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — prostate radiation to 70Gy; nodal radiation to 56Gy

SUMMARY:
The purpose of this study is to examine the clinical feasibility and efficacy of uing IMRT to escalate the biologically effective dose to the pelvic lymph nodes in a short course of radiation therapy. An increased total and biologically effective dose will be delivered to the pelvic lymph nodes (56 Gy at 2 Gy/fraction). The prostate will receive standard "short course" IMRT of radiation (70 Gy at 2.5 Gy/fraction).

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer stage T-T3
* Predicted risk of lymph node involvement > 15%
* Gleason > 7

Exclusion Criteria:

* Distance metastases
* Use of anti-coagulant therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ritter, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University Of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with high-risk prostate adenocarcinoma or radiographic evidence of pelvic lymph node involvement but absence of distal metastases from the Midwest. The last patient completed in February 2016.
Pre-assignment Details: All participants are assigned to the experimental arm.
Groups:
- Experimental: Pelvic nodal and prostatic image-guided IMRT was delivered to high pelvic nodal risk participants to a nodal dose of 56 Gy in 2-Gy fractions with concomitant treatment of the prostate to 70 Gy in 28 fractions of 2.5 Gy
Period: Overall Study
Arm/Group | Experimental
Started | 30
Completed (All participants completed treatment per protocol; 5 died greater than 30 days after last treatment.) | 25
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: Participants with histologically confirmed prostate cancer and no evidence of bone or extrapelvic metastases were enrolled.
Arm/Group | Experimental
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
T stage [Count of Participants; unit: Participants] — Participants with stage T1-T4 disease, as defined by 1997 AJCC classification, were enrolled. The T Stage information of the last 5 participants enrolled is not included. The T stages reported in this table are refer to the following stages:
  T1c: Tumor identified by needle biopsy (eg, because of elevated PSA) T2a: Tumor involves one lobe T2b,c: Tumor involves both lobes T3a,b: Tumor extends through the prostate capsule, extracapsular extension (unilateral or bilateral), and tumor invades seminal vesicle(s) T4: Tumor is fixed or invades adjacent structures other than seminal vesicles
  Participants
    T1c | 9
    T2a | 3
    T2b,c | 7
    T3a,b | 5
    T4 | 1
    Not reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Expected Toxicities
Description: Tolerances to high dose RT to Pelvic Lymph nodes in treatment of prostate cancer; measured by participants experiencing expected toxicities.
Time Frame: Up to 5 years
Population: Only 25 of 30 participants met the minimum follow up thresholds at the time of analysis; the 5 most recently accrued participants' data was not analyzed and is not reflected.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 25
Participants | 13

2. Secondary Outcome: To Evaluate Local Tumor Control and Biochemical Progression-free and Metastasis-free Survival
Description: Clinically evaluate local tumor control and biochemical progression-free and metastasis-free survivals.
Time Frame: 5 years
Population: Data was not collected for this outcome measure. Results can not be reported or analyzed.
Arm/Group | Experimental
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were followed up 1 month upon completion, every 3 months for 1 year after treatment, every 4 months during Years 2 and 3, every 6 months during Years 4 and 5, and then annually, with median follow up time as 25.4 months (range, 4.2 - 57.2 months). Bone scans and CT during follow-ups were not routinely performed but were carried out in the context of rising PSA levels. Of 30 participants, only 25 met the minimum follow up thresholds at the time of analysis.
Description: Toxicity grading is based on a modified RTOG acute/late toxicity grading criteria.
  Serious adverse events are defined as all Grade 4 and Grade 5 toxicities. Acute toxicities are scored from the start of radiation to 90 days after completion of radiation. Late toxicities are scored > 90 days from the completion of radiation therapy for 5 years.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 6/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 13/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=25)
Acute GI Grade 1 (Gastrointestinal disorders) | 13
Acute GI Grade 2 (Gastrointestinal disorders) | 8
Late GI Grade 1 (Gastrointestinal disorders) | 5
Late GI Grade 2 (Gastrointestinal disorders) | 2
Acute GU Grade 1 (Renal and urinary disorders) | 13
Acute GU Grade 2 (Renal and urinary disorders) | 10
Late GU Grade 1 (Renal and urinary disorders) | 9
Late GU Grade 2 (Renal and urinary disorders) | 5
Late GU Grade 3 (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes